CLINICAL TRIAL: NCT07098689
Title: Body Emotional Map Method for the Reduction of Parental Stress Related to Diabetes: a Randomized Study. BEM-02
Brief Title: Body Emotional Map Method for the Reduction of Parental Stress Related to Diabetes
Acronym: BEM-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valentino Cherubini (Other)
Responsible Party: Sponsor-Investigator, Valentino Cherubini, Head of Unit, Paediatric Diabetology Department of Women's and Children's Health "G. Salesi Hospital", AOU OORR Ancona, Via F. Corridoni, 11 60123 Ancona, Italy, Ospedali Riuniti Ancona
Organization: Ospedali Riuniti Ancona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 26072023
Record Dates: First submitted 2025-07-24; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Stress (Psychology); Diabete Type 1
Keywords: BODY EMOTIONAL MAP; PARENTAL STRESS; chronic condition; Type 1 diabetes
MeSH Terms: conditions — Chronic Disease; Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEM group (Experimental): In the BEM group, participants will receive basic information on diabetes management through external resources (medical support, technology, telemedicine, carbohydrate counting techniques) and internal resources (learning effective techniques and behaviors to improve metabolic control).
  Interventions: Other: The BEM (Body Emotional Maps) program
- Control group (Active Comparator): In the control group, basic information on diabetes management will be provided through external resources (medical support, technology, telemedicine, carbohydrate counting techniques) and internal resources (learning effective techniques and behaviors to improve metabolic control).
  Interventions: Other: Control group

INTERVENTIONS:
Other: The BEM (Body Emotional Maps) program — The BEM method involves an intervention with the parents of children with diabetes, conducted in group settings, aimed at facilitating parents' adaptation to their child's "diabetes condition". The BEM method involves an intervention with the parents of children with diabetes, conducted in group settings, aimed at facilitating parents' adaptation to their child's "diabetes condition". The intervention is organized into three sessions.
  The first session consists of an introduction and group formation. The second session involves sharing the onset of diabetes, identifying the most critical daily challenges, and the primary change the participants wish to implement. The third session features the BEM pathway, which includes guided visualization and the creation of a map with spatial anchors.
  Arms: BEM group
Other: Control group — The control group will receive the same diabetes management information, accompanied by parent discussion sessions and recreational activities guided by the diabetes team staff. As with the BEM group, activities will take place over three days in an off-hospital location, in contact with nature.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the impact of the BEM method on stress and well-being in parents of children/adolescents with type 1 diabetes, compared to a standard group approach focused on therapeutic education (control group). The BEM Program involves an experiential, group-based approach facilitated by 2-3 trained facilitators and a maximum of 25 parent participants. Each session takes place over three consecutive days and includes both plenary sessions with the entire group and smaller subgroup activities. Metodology of BEM approach includes: relaxation techniques, breathing exercises, and guided visualizations NLP (Neuro-Linguistic Programming) techniques: spatial anchoring, Time Line therapy, and future pacing. Approaches based on Transactional Analysis (T.A.) and Systemic-Relational frameworks, brief interventions focused on problem-solving. Techniques for enhancing bodily and emotional awareness. Interactive group discussions. The control intervention will take place during a camp specifically dedicated to parents, with the same duration as the BEM program. The intervention includes educational and informational sessions on key aspects of type 1 diabetes management (management of acute complications, importance of glycemic indices, carbohydrate counting, current and emerging perspectives in type 1 diabetes care). In addition, the program includes opportunities for parents to share personal experiences and participate in recreational activities.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children and adolescents under 18 years of age with type 1 diabetes duration exceeding 12 months;
* Parents of children who have never been diagnosed with psychiatric or behavioral disorders;
* Adequate understanding of the Italian language, as assessed by the clinician;
* Parents willing to: Actively participate in group experiential activities; Complete the required questionnaires; Signed informed consent from the participating individual; Signed informed consent for data processing of the minor by both parents (if applicable).

Exclusion Criteria:

Parents:

* with psychiatric conditions
* of patients with psychiatric issues or behavioral disorders
* with any problem that, according to the clinician's judgment, would prevent active participation in group experiential activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Difference in PSI-SF (Parental Stress Index Short-Form) scores after 3 months | From enrollment to 3 months after the participation in the BEM activities
  The primary endpoint is represented by the difference in PSI-SF (Parental Stress Index Short-Form) scores after 3 months of participation in the group activities compared to baseline. PSI-SF subscale scores range from 12 to 60, and the total score from 36 to 180. High subscale scores and a high PSI-SF total score indicate higher levels of stress. Responses above the 85th percentile are considered clinically significant.

SECONDARY OUTCOMES:
Difference in PSI-SF (Parental Stress Index Short-Form) scores after 6 months and in the scores of the individual components of the PSI-SF questionnaire | from enrollment to 6 months from participation in the group activities compared to baseline
  The secondary endpoint is represented by the difference in PSI-SF (Parental Stress Index Short-Form) scores (total and of each suscale) after 6 months of participation in the group activities compared to baseline. Subscale scores range from 12 to 60, and the total score from 36 to 180. High subscale scores and a high PSI-SF total score indicate higher levels of stress. Responses above the 85th percentile are considered clinically significant.
Patient Health Questionnaire (PHQ-9) | From enrollment to 3 and 6 months from participation in the group activities compared to baseline
  Difference in the scores of the Patient Health Questionnaire (PHQ-9) for the assessment of depression and depressive symptoms after 3 and 6 months from the baseline. Each symptom is rated on a 4-point scale. Scores range from 0 to 27, with different levels of depression severity depending on the score: 10-14 = Mild major depression; 15-19 = Moderate major depression; ≥ 20 = Severe major depression.
General Anxiety Disorder (GAD-7) | From enrollment to 3 and 6 months from participation in the group activities compared to baseline.
  Difference in the scores of the General Anxiety Disorder (GAD-7) questionnaire for the assessment of anxiety and anxious symptoms. Scores of 0, 1, 2, or 3 are assigned for symptoms occurring "not at all," "several days," "more than half the days," and "almost every day," respectively. The scores are then summed and range from 0 to 21. Scores of 5, 10, and 15 represent cutoffs for mild, moderate, and severe anxiety, respectively.
Brief Pittsburgh Sleep Quality Index (B-PSQI) | From enrollment to 3 and 6 months from participation in the group activities compared to baseline
  Difference in the scores of the Brief Pittsburgh Sleep Quality Index (B-PSQI) for the assessment of sleep disturbances. For each area, a score from 0 (highest positive) to 3 (lowest negative) is assigned, as follows: "Never during the last month" = 0; "Less than once a week" = 1; "1 or 2 times a week" = 2; "3 or more times a week" = 3. Summary score is then generated, obtained by adding the scores for the individual areas, with a value ranging from 0 to 21. Score between 5 and 7 indicates mild sleep disturbances may occur; score above 7 indicates that it is recommended to consult a doctor for a more in-depth evaluation of sleep disturbances.
Parental Self-Efficacy for the Management of Diabetes Mellitus (PSESDM) questionnaire. | From enrollment to 3 and 6 months from participation in the group activities compared to baseline
  Difference in the scores of the Parental Self-Efficacy for the Management of Diabetes Mellitus (PSESDM) questionnaire for the evaluation of self-efficacy perception in managing their child's diabetes. Responses range from 1 = "Strongly disagree" to 5 = "Strongly agree." Items 1, 2, 6, and 7 are reverse-scored. The total score on the measure ranges from 8 to 40. A higher score on the PSESDM represents greater parental confidence in managing their child's diabetes.
Coping Orientation to the Problems Experienced - Italian Version (COPE-NVI) | From enrollment to 3 and 6 months from participation in the group activities compared to baseline
  Difference in the scores of the Coping Orientation to the Problems Experienced - Italian Version (COPE-NVI) questionnaire for assessing parental adaptation and coping strategies. Responses to each question are given on a scale from 1 = "I usually don't do it" to 4 = "I almost always do it." Individual question scores are summed separately for each of the 5 areas.
Glucometric data of children/adolescents | From enrollment to 3 and 6 months from participation in the group activities compared to baseline.
  Difference in glucometric data of children/adolescents:
  * HbA1c; if CGM, glucose values in the last 15 days:
  * Time in Range;
  * Time below range level 1;
  * Time below range level 2;
  * Time above range level 1;
  * Time above range level 2,
  * Average blood glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Women's and Children's Health Azienda Ospedaliero Universitaria delle Marche, G. Salesi Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT07098689/Prot_000.pdf